CLINICAL TRIAL: NCT04692701
Title: Pulvinar Stimulation in Epilepsy: a Pilot Study
Acronym: PULSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-49; 2020-A02119-30 (Other: ID RCB)
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Epilepsy
Keywords: epilepsy; pulvinar; seizures; deep brain stimulation
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulvinar stimulation (Experimental): Medial pulvinar deep brain stimulation
  Interventions: Device: Pulvinar deep brain stimulation

INTERVENTIONS:
Device: Pulvinar deep brain stimulation — Stimulation of the medial pulvinar

SUMMARY:
Deep brain stimulation (DBS) is one of the neuromodulation techniques that can be indicated in patients suffering from refractory epilepsies, especially when an open resection has failed or is not indicated, and vagal nerve stimulation (VNS) demonstrated no efficacy. Benefits such as reduction of seizure frequency have been shown for thalamic stimulation of the anterior thalamic nucleus (ANT), however it has limited efficacy and non-optimal neurocognitive outcome, making the search for other targets crucial in this context. We propose a novel target for DBS stimulation in drug-resistant epilepsy namely the medial pulvinar thalamic nucleus (PuM).

This target has been chosen based on previous retrospective studies demonstrating that PuM is involved during focal seizures and in loss of consciousness and seizure termination. PuM stimulation also showed potential encouraging results based on the feasibility and safetu studies recently published.

The main objective is to obtain a significant percentage of seizure reduction after 12 months of PuM stimulation compared to baseline period. Quality of life and the relationship with psychiatric and cognitive comorbidities will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 60 years old
* Focal or multifocal drug-resistant epilepsy not operable or failure of epilepsy surgery
* Vagal nerve stimulation failure (after at least 1 year of treatment or stopped early for worsening seizures)
* Either patients with epilepsy whose characteristics suggest that it may respond better to stimulation of the pulvinar than the anterior thalamic nucleus stimulation (i.e. posterior quadrant epilepsy, motor/premotor epilepsy, operculo-insular epilepsy, temporal plus epilepsy, lateral temporal epilepsy) or/and patients with previous anterior thalamic nucleus stimulation failure (after 2 years of treatment or stopped early for worsening seizures)
* Number of seizures > 4 / month during the baseline (3 months) and before the V0 for at least 3 months
* Total IQ > 55
* Give written consent to the study after receiving clear information
* Be a beneficiary or affiliated to a health insurance plan
* For women of childbearing potential, a pregnancy test must be negative before inclusion.

Exclusion Criteria:

* Difficulty to read or understand the French language, or inability to understand the information regarding the study.
* Generalized epilepsy
* Presenting contraindication to MRI, a serious intercurrent pathology, a progressive brain tumor.
* Pregnancy or breastfeeding
* Present a history of attempted suicide in the 6 months prior to inclusion or a score ≥ 2 in item 10 of the Montgomery and Asberg Depression Scale (MADRS).
* Present a surgical or anaesthetic contraindication.
* Require long-term anticoagulant or platelet aggregation therapy.
* Hereditary bleeding disorders of coagulation
* Non obliterated AVM
* History of Herpes virus brain infection
* Total IQ below 55.
* Patients with less than 4 seizures a month
* To be hospitalized under duress (HO / HDT)
* Major under guardianship or curatorship
* Person deprived of liberty by judicial decision
* Patient currently participating in another clinical trial or having participated in a clinical trial in the month prior to inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Number of seizures | Change from baseline to 12 months
  Events will be recorded using a seizure diary

SECONDARY OUTCOMES:
Score of depression | Change from baseline to 12 months
  NDDI-E
Score of anxiety | Change from baseline to 12 months
  GAD-7
Score of quality of life | Change from baseline to 12 months
  QOLIE
Score of epilepsy severity | Change from baseline to 12 months
  Chalfont

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier Arnaud, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Service de Neurologie, Nice, France, France

IPD SHARING:
Plan to Share IPD: No